CLINICAL TRIAL: NCT00435721
Title: The Families Coping With Mental Illness Program
Brief Title: Families Coping With Mental Illness Program
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: North Suffolk Mental Health Association (Other)
Collaborators: Mclean Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: CORRC 03-2003
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2007-02-15 (Estimated); Status verified 2007-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; family psychoeducation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

INTERVENTIONS:
Behavioral: Psychoeducation

SUMMARY:
The current study aims to develop and evaluate a practical, short-term support and education program for relatives of individuals with schizophrenia. This program has been developed to maximize efficiency and effectiveness in the following ways:

1. The intervention specifically targets those factors empirically demonstrated to improve family functioning and well being. Specifically, this pilot intervention aims to: a) increase relatives' knowledge about schizophrenia spectrum disorders; b) help families attribute distressing behaviors of their ill relatives more accurately, by helping them to distinguish behaviors that are directly related to the illness from personality characteristics; c) improve attitudes towards the patient and reduce stress in interactions with the patient; d) encourage problem-focused coping strategies; e) reduce burden; f) provide opportunities for relatives to expand their social support network; g) help families learn about and utilize community resources.
2. The program involves both individual and multifamily group components, in order to reap the benefits of both formats. Specifically, multifamily psychoeducation groups (involving individuals from several different families) tend to be more economical and allow participants to learn from each other, increase their social support networks, and reduce feelings of stigma. In contrast, individualized programs can target the specific needs of participants.

DETAILED DESCRIPTION:
Format of intervention:

The program contains the following components:

Four multiple family group sessions:

* Session 1: Understanding the illness
* Session 2: Treatments and community resources
* Session 3: Coping with the illness
* Session 4: Reducing stress in the family

  2. Two individual consultation sessions with the group leader (occurring before and after the group) The principal investigator will conduct all group and individual sessions. Since the intervention is brief, emphasis is placed on introducing concepts and helping relatives learn how to obtain more information for themselves, rather than on practicing and adopting all skills that are introduced. Materials are provided to read between sessions to supplement the didactic presentations and allow maximum time for relatives to discuss how topics relate to their personal experiences. In addition, group members are asked each week to report on how they applied strategies discussed in the group and whether or not they found them to be effective.

Subjects:

The participants in this study will be a minimum of 50 adult relatives of individuals with schizophrenia or schizoaffective disorder. Up to three relatives per family may participate in the program. Groups will contain between 4 and 10 people from a minimum of three families.

Procedure:

Assessments, consultations, and groups will take place at McLean Hospital or the Freedom Trail Clinic to prevent external environmental influences from affecting data collection and to ensure that the interviews will be held in a confidential location. A wait-list control design will be used to evaluate the efficacy of this intervention. Clients will be assessed initially on a number of dimensions (specified below) by a trained, reliable research assistant. These clients will be randomly assigned to either an intervention (psychoeducation right away) or a wait-list control condition . The psychoeducation program will consist of four weekly, 2 ½ -hour multifamily group sessions and two individualized pre- and post-group consultation sessions. Clients in the control condition will receive psychoeducation after the intervention group has completed the program. Upon completion of the psychoeducation program, a research assistant will re-evaluate relatives in both the intervention and the wait-list control group. To minimize interviewer bias, this research assistant will be blind to which condition (intervention or wait-list) the clients were assigned.

Measures:

Self-report instruments and audiotaped structured interviews included in the pre- and post-intervention assessments will measure knowledge about schizophrenia, coping strategies, perceived burden, expressed emotion, attribution of illness symptoms and behaviors, quality and use of social support network, and depression and anxiety among participants. Participants will also be asked to provide demographic information such as age, ethnicity, socioeconomic status, relationship to patient (e.g., parent, sibling), and living situation (whether or not participant resides with patient). Participants who do not live with patients will be asked to identify the number of hours per week spent in caregiving activities (e.g., assistance with activities of daily living or providing companionship). In addition, the post-intervention assessment will include some measures of client satisfaction. (Copies of all measures are attached).

Specific hypothesis:

Compared to wait list control subjects, subjects who have participated in the intervention will show decreased levels of perceived burden, depression, anxiety, high expressed emotion, and attributions of control. Furthermore, they will exhibit increased knowledge regarding the illness, use of community resources, and perceived social support.

10. Duration of the study and the subject's involvement in the study: Subject participation in this study will be approximately 6 weeks for the intervention group and 12 weeks for the wait list group. Subjects in the intervention group will come to McLean 6 times (two interview and consultation sessions and four educational sessions). Subjects in the wait list group will come to McLean 7 times (this includes one additional interview session after the wait list period, before starting the group). The duration of the study is expected to be at least 1 year. We would like to continue recruiting subjects until a least 50 subjects have participated.

ELIGIBILITY:
Inclusion Criteria:

* Self identified family members of individuals with schizophrenia or schizoaffective disorder or psychosis NOS
* 18 years old or over

Exclusion Criteria:

* Own diagnosis of schizophrenia /schizoaffective disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-06; Study Completion 2005-08

PRIMARY OUTCOMES:
Family knowledge
Family Burden
Expressed emotion

SECONDARY OUTCOMES:
Social Support
Coping Strategies
Confidence in knowledge
Use of community resources

CONTACTS AND LOCATIONS:
Overall Officials: Michelle S. Friedman-Yakoobian, Ph.D., Principal Investigator — Massachusetts General Hospital, Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - McLean Hospital, Belmont, Massachusetts
  - Freedom Trail Clinic North Suffolk Mental Health Association, Boston, Massachusetts